CLINICAL TRIAL: NCT02346006
Title: CHAMPS Eye Study - Myopia and Retinal Vascular Geometry in Relation to Physical Activity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Kristian Lundberg, MD, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CES 001
Record Dates: First submitted 2015-01-09; First posted 2015-01-26 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Child; Motor Activity; Myopia
Keywords: Exercise; Visual Acuity; Blood Vessels; Retina; Choroid
MeSH Terms: conditions — Motor Activity; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Physical activity (Experimental): Subject from schools with more physical activity.
  Interventions: Behavioral: More physical activity.

INTERVENTIONS:
Behavioral: More physical activity. — Subjects receiving more physical activity in school.

SUMMARY:
An increasingly physical inactive lifestyle in the Western World has led to a higher number of lifestyle -related diseases. The consequences are now already present in childhood with an increased prevalence of overweight, obesity, and diabetes. Inactivity is also accompanied by cardiovascular iseases and is also thought to be associated with an increased incidence of nearsightedness (myopia).

Myopia is the most frequent eye disease globally, and causes severe personal and societal expenses and may additionally lead to secondary eye disorders such as retinal detachment, glaucoma, and cataract.

The retina is the only place in the human body where it is possible to directly inspect the blood vessels (microvasculature). Photography of the eye background allows a noninvasive examination of the retinal structure in which it is possible to make measurements on the retinal blood vessels.

It is well known that early vascular chances can be detected with this method and that there are correlation between these changes and systemic diseases, such as hypertension, stroke and other cardiovascular diseases.

This study is a new subproject in The Childhood Health, Activity, and Motor Performance School (CHAMPS) Study Denmark, also known as the Svendborg Project. The project has a well-defined cohort with originally 1515 school students who since 2007 have been divided into two groups: schools with extra exercise during school hours and matched traditional schools. CHAMPS-DK aims to investigate the effect of increased physical activity on current and future health of children and adolescents.

Thanks to this unique child cohort it is possible to investigate the correlation between physical activity, myopia and retinal vascular diameters in a large group of Danish schoolchildren. We want to study the degree and reversibility of physical activity and its effect on the development of myopia and retinal blood vessel changes. However, there is still a lack of knowledge about the correlation between physical activity and retinal vascular diameters in children. Furthermore, it is still unclear whether physical activity can prevent the development of myopia; such a realization could have far-reaching consequences in form of a modified approach to the necessity for exercise and, furthermore, potentially a significant socio-economic benefit.

DETAILED DESCRIPTION:
Introduction Increasingly physical inactive lifestyle in the western world has led to an increase in life style related diseases. The consequences are now already present in childhood with an increased prevalence of overweight, obesity and diabetes. Inactivity is also accompanied by cardiovascular diseases and is also thought to be associated with an increased incidence of near sightedness (myopia).

Myopia is the world's most occurring eye disease, and is usually caused by increasing length growth of the eye. Myopia in itself leads to great personal and societal costs and in addition it also lead to secondary eye disorders such as retinal detachment, glaucoma and cataract. The growth of the eye length is principally developed until mid-childhood, witch is why it is these years witch is most valuable to investigate the underlying factors of the development of myopia.

The prevalence of myopia has increased significantly the recent decades, without a known cause. Particularly in Asia, there has been a very high and dramatically increasing prevalence of myopia - in some urbanized areas up to 80-90% among children in the final year of primary school people.

Myopia is caused by a combination of genetic and environmental factors. Lifestyle changes such as reduced physical activity and more close-up work is thought to of great importance.4 Conversely, there is also evidence of a possible protective effect of outdoor presence in the development of myopia. We do not kwow if the protective effect is due to the total time spent outdoors per se or the increased physical activity, although a small study describe a slower development and lower degrees of myopia in children who used more time on outdoor activities and sports than children in a control group. In addition a Danish study of college students (physical education students -vs. medical students) found an association between physical activity, student activity and myopia suggesting a preventive effect of physical activity and less intense study activity on the development and progression of myopia.

It is still unclear whether physical activity can prevent the development of myopia - a such realization could have far-reaching consequences in form of a modified approach to the necessity for exercise and a consequent significant socio-economic benefit.

The retina is the only place in the human body where it is possible to directly inspect the microvasculature. Photography of the eye background (fundus photography) is a non-invasive examination of the retinal structure in which it is possible to make measurements on the retinal blood vessels. Semi automated measurements of retinal vascular diameters is a simple and validated method to examine the retinal system.

Several large studies have shown a correlation between retinal vessel diameters and systemic diseases such as hypertension, stroke and other cardiovascular diseases in adults. Furthermore, studies also demonstrate retinal vascular changes in children comparable to the changes in adults , including thinner retinal arteries in children with hypertension.

Blood pressure levels are significantly increased among children and adolescents over the last ten years, which can be related to an increase in obesity. There is also a correlation between a physically inactive lifestyle and obesity. High blood pressure in children and adolescence leads to increased risk of cardiovascular disease risk later on in life , including the development of early atherosclerosis .

There is still missing considerable knowledge about the correlation between physical activity and retinal vascular diameters in children. By being able to identify retinal vessel diameters as a risk factor marker for later development of cardiovascular disease, it will be possible at an early stage to identify those children who will benefit from targeted preventional efforts.

Using a unique child cohort we want to investigate the correlation between physical activity, myopia and retinal vascular diameters in a large group of Danish schoolchildren. We will study the degree and reversibility of physical activity and its effect in the development of myopia and retinal vasculopathy.

The study - material The current study is a new subproject in The Childhood Health, Activity, and Motor Performance School (CHAMPS) Study Denmark. CHAMPS-DK aims to investigate the effect of increased physical activity on current and future health of children and adolescents.

In 2007, the city council in Svendborg took the decision to provide increased levels of suitable physical activities in some of their primary schools, with the aim to improve the physical health of children. Before starting the Svendborg Project, all 19 primary schools in Svendborg were invited, of which six choose to participate. A committee consisting of school principals and physical education teachers from these schools made a proposal based on Team Denmark training concept for children.

The project has a well-defined cohort with originally 1515 school students who since 2007 has been divided into two groups: 775 in the six schools with extra exercise during school hours and 750 in six matched traditional schools. The six sports schools introduced 6 hours of sport per week versus a normal hour for sport at 2 hours a week.

Students have so far been followed for six years and researchers from Hans Christian Andersen Children's Hospital, University Hospital and Centre of Research in Childhood Health (RICH), SDU has studied the effect of physical activity on lifestyle diseases, back problems, sports injuries, etc.

Students - initially aged 6 to 10 years - are followed and studied in a variety of areas. At baseline were made surveys, demographic data collected, objective tests, physical and biological tests, including DEXA scans and blood tests. In addition, visual data on each student from healthcare study at school start are noted, so that it possible to determine who was myopic at that time.

Each week throughout the study period, students and parents answered a text message with questions about the student's leisure- and sports activities, duration and type, and whether any problems encountered in the musculoskeletal system. In addition, twice a year, data on health habits, physical objective measures, balance, endurance capacity, bone status, lifestyle diseases, injuries and musculoskeletal problems has been collected.

For some periods students are equipped with an accelerometer - a device that can objectively measure the amount and degree of physical activity. With data collection from the weekly SMS updates and continuous measurements with the accelerometer, it is possible all the time to know each student's precise level of exercise and have a detailed knowledge of the student's physical form.18,

Purpose The project serves to investigate the effect physical activity has on 1) the development of myopia and 2) the retinal vascular geometry, including whether the latter can be used as a marker for cardiovascular risk in children.

With this project, we also strive to promote research cooperation across the departments at Odense University Hospital and the Research Unit of Ophthalmology, Institute of Clinical Research and RICH.

Hypothesis

We expect that physical activity has a protective effect against myopia as well as retinal vasculopathy and make the following hypothesis:

1. Physical activity - especially outdoor activity - is associated with less myopia in children of school age
2. Physical activity is associated with more optimal retinal vascular diameters and therefore a more favourable cardiovascular risk profile.

Method

1. The study is conducted as a cross-sectional study aimed to associate the current level of physical activity (assessed by self-report and accelerometer) with 1) the degree of myopia and 2) the retinal vascular diameters.
2. The study will also be a follow-up of the baseline data collected from the cohort at school start, where school nurse measurements (and later reference to practicing ophthalmologists) has been possible to identify students who was already myopic. This makes it possible to create a longitudinal assessment of the degree of myopia in the study.

Data collection

In the spring 2015, 700 of the enrolled students (currently in 7th-10th grade) in the CHAMPS study will be called for examination at Odense University Hospital, where the following data is collected:

Non ophthalmological data:

Age, sex, weight, height, cardiovascular risk factors (lipid status, DEXA scans, vitamin D), physical status and outdoor level (assessed from type of school, SMS reporting and accelerometer).

Ophthalmological data:

Visus (ETDRS), autorefraction in cycloplegia, refractional status (axis length, k-number), tonometry, fundus photography (vascular diameter) and spectral-domain optical koherens tomography (SD-OCT).

Analysis and data processing In the study retinal photographs and OCT are recorded a fundus camera (Topcon 3D OCT, Tokyo, Japan). To measure and analyse the retinal vessels a semi-automated computer program (IVAN) is used. It can give numerous information and calculate the diameters of arterioles and venules.

Power calculation The study will have a fixed cohort of 700 students. In order to ensure that there is enough power to investigate the anticipated correlations, the following power calculations are made (SigmaPlot, version 12, Systat Software Inc., San Jose, California, United States).

Visus: Requires the inclusion of at least 64 students in order to detect a difference of 5 ETDRS letters with the following assumptions: normal distribution, statistical power: 80% significance level (α): 5%, standard deviation (SD): 10 ETDRS letters.

Refraction: Requires the inclusion of at least 194 students to detect a difference 0.50 diopter (power: 80%, α = 5%, SD = 1.75D).

Arteriolar vascular diameter: Requires the inclusion of at least 125 students to detect a change of 5 microns (power: 80%, α: 5%, SD = 14 microns).

Overall the cohort meets the requirements.

Perspectives The study may later form the basis for a follow-up study in which the present investigations may constitute the baseline data for a longitudinal study to investigate 1) the role of physical activity in the final development of myopia in the cohort and 2) the correlation of retinal vascular diameter status to later development of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Children from the The Childhood Health, Activity, and Motor Performance School Study Denmark (The CHAMPS-study DK) cohord.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Myopic status in relation to physical activity (longitudinal data on physical activity) | 7 years
  Myopic status in relation to longitudinal data on physical activity

SECONDARY OUTCOMES:
Retinal vessel geometry (caliber) | None (analyzes on data from tests in march to july 2015, 4 months)
  Cross-sectional results.
  Change in vessel geometry:
  Caliber: Using computerised software - IVAN.
Choroidal thickness | None (analyzes on data from tests in march to july 2015, 4 months)
  Cross-sectional results. Using Enhanced Depth Imaging Spectral Domain Optical Coherence Tomography
Myopic status (data from tests in spring 2015) | None (analyzes on data from tests in march to july 2015, 4 months)
  Cross-sectional results
Myopia development | 10 years. Changes from baseline.
  Cross-sectional results compared with date from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Lundberg, MD, Principal Investigator — Department of Ophthalmology, Odense University Hospital

REFERENCES:
- [Background] Andersen LB, Wedderkopp N, Hansen HS, Cooper AR, Froberg K. Biological cardiovascular risk factors cluster in Danish children and adolescents: the European Youth Heart Study. Prev Med. 2003 Oct;37(4):363-7. doi: 10.1016/s0091-7435(03)00145-2. PMID 14507494
- [Background] Parssinen O, Leskinen AL, Era P, Heikkinen E. Myopia, use of eyes, and living habits among men aged 33-37 years. Acta Ophthalmol (Copenh). 1985 Aug;63(4):395-400. doi: 10.1111/j.1755-3768.1985.tb01551.x. PMID 4050359
- [Background] Angle J, Wissmann DA. The epidemiology of myopia. Am J Epidemiol. 1980 Feb;111(2):220-8. doi: 10.1093/oxfordjournals.aje.a112889. PMID 7355884
- [Background] Morgan IG, Ohno-Matsui K, Saw SM. Myopia. Lancet. 2012 May 5;379(9827):1739-48. doi: 10.1016/S0140-6736(12)60272-4. PMID 22559900
- [Background] Lin LL, Shih YF, Hsiao CK, Chen CJ. Prevalence of myopia in Taiwanese schoolchildren: 1983 to 2000. Ann Acad Med Singap. 2004 Jan;33(1):27-33. PMID 15008558
- [Background] He M, Zeng J, Liu Y, Xu J, Pokharel GP, Ellwein LB. Refractive error and visual impairment in urban children in southern china. Invest Ophthalmol Vis Sci. 2004 Mar;45(3):793-9. doi: 10.1167/iovs.03-1051. PMID 14985292
- [Background] Saw SM, Chua WH, Wu HM, Yap E, Chia KS, Stone RA. Myopia: gene-environment interaction. Ann Acad Med Singap. 2000 May;29(3):290-7. PMID 10976381
- [Background] Rose KA, Morgan IG, Ip J, Kifley A, Huynh S, Smith W, Mitchell P. Outdoor activity reduces the prevalence of myopia in children. Ophthalmology. 2008 Aug;115(8):1279-85. doi: 10.1016/j.ophtha.2007.12.019. Epub 2008 Feb 21. PMID 18294691
- [Background] Parssinen O, Lyyra AL. Myopia and myopic progression among schoolchildren: a three-year follow-up study. Invest Ophthalmol Vis Sci. 1993 Aug;34(9):2794-802. PMID 8344801
- [Background] Jacobsen N, Jensen H, Goldschmidt E. Does the level of physical activity in university students influence development and progression of myopia?--a 2-year prospective cohort study. Invest Ophthalmol Vis Sci. 2008 Apr;49(4):1322-7. doi: 10.1167/iovs.07-1144. PMID 18385044
- [Background] Cheung CY, Ikram MK, Sabanayagam C, Wong TY. Retinal microvasculature as a model to study the manifestations of hypertension. Hypertension. 2012 Nov;60(5):1094-103. doi: 10.1161/HYPERTENSIONAHA.111.189142. Epub 2012 Oct 8. PMID 23045470
- [Background] Grauslund J, Hodgson L, Kawasaki R, Green A, Sjolie AK, Wong TY. Retinal vessel calibre and micro- and macrovascular complications in type 1 diabetes. Diabetologia. 2009 Oct;52(10):2213-7. doi: 10.1007/s00125-009-1459-8. Epub 2009 Jul 18. PMID 19618163
- [Background] Hanssen H, Siegrist M, Neidig M, Renner A, Birzele P, Siclovan A, Blume K, Lammel C, Haller B, Schmidt-Trucksass A, Halle M. Retinal vessel diameter, obesity and metabolic risk factors in school children (JuvenTUM 3). Atherosclerosis. 2012 Mar;221(1):242-8. doi: 10.1016/j.atherosclerosis.2011.12.029. Epub 2011 Dec 27. PMID 22244041
- [Background] Gopinath B, Baur LA, Wang JJ, Teber E, Liew G, Cheung N, Wong TY, Mitchell P. Blood pressure is associated with retinal vessel signs in preadolescent children. J Hypertens. 2010 Jul;28(7):1406-12. doi: 10.1097/HJH.0b013e3283395223. PMID 20410837
- [Background] Muntner P, He J, Cutler JA, Wildman RP, Whelton PK. Trends in blood pressure among children and adolescents. JAMA. 2004 May 5;291(17):2107-13. doi: 10.1001/jama.291.17.2107. PMID 15126439
- [Background] Raitakari OT, Juonala M, Kahonen M, Taittonen L, Laitinen T, Maki-Torkko N, Jarvisalo MJ, Uhari M, Jokinen E, Ronnemaa T, Akerblom HK, Viikari JS. Cardiovascular risk factors in childhood and carotid artery intima-media thickness in adulthood: the Cardiovascular Risk in Young Finns Study. JAMA. 2003 Nov 5;290(17):2277-83. doi: 10.1001/jama.290.17.2277. PMID 14600186
- [Background] Berenson GS, Srinivasan SR, Bao W, Newman WP 3rd, Tracy RE, Wattigney WA. Association between multiple cardiovascular risk factors and atherosclerosis in children and young adults. The Bogalusa Heart Study. N Engl J Med. 1998 Jun 4;338(23):1650-6. doi: 10.1056/NEJM199806043382302. PMID 9614255
- [Background] Wedderkopp N, Jespersen E, Franz C, Klakk H, Heidemann M, Christiansen C, Moller NC, Leboeuf-Yde C. Study protocol. The Childhood Health, Activity, and Motor Performance School Study Denmark (The CHAMPS-study DK). BMC Pediatr. 2012 Aug 20;12:128. doi: 10.1186/1471-2431-12-128. PMID 22906115
- [Background] Heidemann M, Molgaard C, Husby S, Schou AJ, Klakk H, Moller NC, Holst R, Wedderkopp N. The intensity of physical activity influences bone mineral accrual in childhood: the childhood health, activity and motor performance school (the CHAMPS) study, Denmark. BMC Pediatr. 2013 Mar 2;13:32. doi: 10.1186/1471-2431-13-32. PMID 23452342
- [Background] Lundberg K, Kawasaki R, Sjolie AK, Wong TY, Grauslund J. Localized changes in retinal vessel caliber after focal/grid laser treatment in patients with diabetic macular edema: a measure of treatment response? Retina. 2013 Nov-Dec;33(10):2089-95. doi: 10.1097/IAE.0b013e3182891dda. PMID 23514802